CLINICAL TRIAL: NCT07006649
Title: CHOPXE - Analysis of Choriocapillaris Flow Deficits in Patients With Pseudoxanthoma Elasticum
Acronym: CHOPXE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC24_0254; 2025-A00674-45 (Other: ANSM (French Ministry of Health))
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pseudoxanthoma Elasticum; Tomography, Optical Coherence; Retinal Disease
Keywords: comparative studies; observational study; adult; cross-sectional studies; healthy volunteers
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers arm with opthtalmologic evaluation (Experimental)
  Interventions: Diagnostic Test: Opthtalmologic diagnosis tests

INTERVENTIONS:
Diagnostic Test: Opthtalmologic diagnosis tests — Volunteer will be tested with : measurement of visual acuity, slit-lamp examination, fundus examination, optical coherence tomography

SUMMARY:
This observational study sets out to compare choriocapillaris flow deficits between healthy control subjects and patients with pseudoxanthoma elasticum. Pseudoxanthoma elasticum (PXE) is a rare, incurable hereditary disease caused by genetic mutations. The condition is characterised by excessive tissue mineralisation, which can result in a range of dermatological, vascular, and ophthalmological complications. Among these complications is the potential for visual impairment. The management of this condition is focused on the treatment of its complications. Degeneration of the retina and the choroid (the layer responsible for ensuring its vascularisation) occurs in the eye, resulting in premature degeneration. We would like to study the premature alteration of these structures, which could subsequently be used as an objective marker of the evolution of pseudoxanthoma elasticum.

DETAILED DESCRIPTION:
CHOPXE is a single-center, cas-control, cross-sectional study with the objective of comparing choriocapillaris flow deficits by OCT angiography (OCT-A) between healthy control subjects and patients with pseudoxanthoma elasticum.

Study rationale Pseudoxanthoma elasticum (PXE) is a rare disorder, affecting between 1 in 25,000 and 1 in 100,000 people. This autosomal recessive disorder is caused by mutations in the ABCC6 gene. Mutations in the ABCC6 gene have been demonstrated to impair cellular efflux of ATP, which is ordinarily converted to inorganic pyrophosphate (PPi) and adenosine. PPi is a potent endogenous inhibitor of calcification, while adenosine contributes indirectly to calcification inhibition by suppressing the synthesis of tissue-nonspecific alkaline phosphatase (TNAP).

The disease has been shown to cause ectopic mineralization and fragmentation of tissue elastic fibres.

* The initial indications of the disease manifesting in the skin are frequently observed in childhood or adolescence. These initial signs evolve slowly and unpredictably, as evidenced by the appearance of papular skin lesions in flexural zones.
* The ophthalmological manifestations (peau d'orange, angioid striae, sub-retinal neovascularization, optic nerve drusen) may be responsible for visual impairment through central blindness.
* The presence of vascular manifestations, including peripheral arterial disease, gastrointestinal bleeding and ischaemic stroke, has been identified as a contributing factor to the premature mortality observed in patients with PXE, when compared to the general population.

Angers University Hospital is a national rare diseases reference center for PXE, with an active file of nearly 300 patients.

At present, there is no treatment available for pseudoxanthoma elasticum, with the exception of treatment for complications. A number of treatments are currently under investigation; however, there is an absence of relevant objective criteria with which to evaluate their efficacy.

The wall of the eyeball is composed of three tunics: the sclera, the choroid and the retina. The retina is composed of multiple layers, with the deepest layer being the retinal pigment epithelium (RPE). The choriocapillaris constitutes the most superficial layer of the choroid, providing blood supply to the outer retina and photoreceptors. The existence of a mutual dependence between these two structures has been established; the choriocapillaris requires the regulatory factors (vascular endothelial growth factor inhibitors) secreted by the RPE for its functionality. Conversely, the RPE is dependent on nutrients and oxygen from the systemic circulation via the choriocapillaris bloodstream to supply the photoreceptors.

Bruch's membrane is a structure located between the retinal pigment epithelium and the choriocapillaris (between the neuroretina and the systemic circulation), which regulates the exchange of molecules between these tissues. The process of pathological mineralization in pseudoxanthoma elasticum has been demonstrated to induce alterations in the exchange mechanisms between these structures, which may potentially result in the premature degradation of photoreceptors and the choriocapillaris.

Optical coherence tomography (OCT) is a widely utilised diagnostic tool in ophthalmology consultations, enabling precise analysis of retinal structures and the optic nerve. This advanced technology boasts a resolution of up to the micrometer, with no need for contact with the eye and a non-invasive procedure. This is an optical ultrasound mode, based on light interferometry. The technology utilises laser reflection from various anatomical structures to facilitate the measurement of retinal thickness. In 2014, a new imaging technology for the retinal and choroidal vascular network was developed from OCT: OCT angiography (OCT-A). The technology is based on the principle of detecting the movements of diffracting particles, such as red blood cells, in sequential OCT B-scans taken at the same point on the retina several times. This makes it possible to objectify the presence of blood vessels. The advent of this new examination has facilitated the analysis of retinal and choroidal vascularization, and in particular retinal and choroidal microcirculation in vivo, such as the choriocapillaris, on a routine clinical basis, which had previously been inaccessible.

Consequently, numerous researchers have initiated studies of the choriocapillaris, with a particular focus on the flow deficits of the choriocapillaris. This is due to the fact that the lateral resolution of OCT-A is approximately equivalent to the macular intercapillary distance, thereby precluding direct observation of the vascularization of the choriocapillaris. The choriocapillaris is responsible for relaying the systemic circulation to the outer retina, thereby providing nutrients and oxygen to the photoreceptors. Consequently, impairment to the choriocapillaris could potentially play a pivotal role in the development of numerous retinal pathologies.

A first study revealed the presence of choriocapillary flow deficits in patients exhibiting angioid streaks on the fundus, including two patients with PXE. These findings were subsequently corroborated by a subsequent study conducted on 21 patients with PXE in the pre-atrophic stages. These results, if confirmed by further studies on larger samples, could make it possible both to use choriocapillary flow deficits for the early diagnosis of PXE, as an additional diagnostic argument in atypical cases, but also to serve as an objective and relevant biomarker for interventional studies evaluating the efficacy of treatment under development.

Patient recruitment The selection of healthy control subjects is made from the database of healthy volunteers at the Clinical Research Centre (CRC) of Angers University Hospital (France), who meet the eligibility criteria. In addition, this study may also be offered to eligible persons waiting for a consultation or accompanying a relative in Angers University Hospital Ophthalmology Department.

The planned inclusion period is 1 year. PXE patients whose data will be used for matching have already been recruited as part of routine care.

It is anticipated that the study will encompass a total of 60 healthy control subjects and 60 PXE patients.

Data collected Following inclusion, participants' characteristics are collected (age, sex, general history, ophthalmological history, cardiovascular events, whether or not digestive bleeding has occurred, and whether antiaggregant or antiplatelet therapy is being taken).

The ophthalmological assessment is carried out during a scheduled consultation at the Angers University Hospital Ophthalmology Department. It includes a measurement of best corrected visual acuity, a slit lamp examination, a fundus and an OCT-A scan. These elements enable us to rule out ophthalmological pathology (maculopathy, retinopathy, optic neuropathy, glaucoma).

If the quality of the OCT-A signal is unsatisfactory (too much artifact and/or image quality signal less than 50/100), the participant is offered pupillary dilatation if there is no contraindication to dilatation (risk of closure of the iridocorneal angle). Dilatation is performed by instilling tropicamide into both eyes.

For PXE patients, additional data of interest (described below) are collected from the patient's medical file.

* ABCC6 gene mutations
* Presence or absence of disease-specific dermatological changes
* Presence or absence of disease-specific ophthalmological changes
* Presence or absence of inflammatory skin flares
* Presence or absence of arterial stenosis of the lower limbs
* Presence or absence of carotid artery dysplasia We also collect patients' age and weight, in order to calculate their body mass index and the presence of cardiovascular risk factors (diabetes, hypertension, smoking, dyslipidemia), as these factors can influence choriocapillary flow deficits, and will enable us to compare the characteristics of patients and controls.

For both PXE patients and healthy subjects, we will select a single eye for our study, choosing the eye with the least choriocapillaris flow deficits (lowest mean percentage on 6x6mm sections).

The OCT-A choriocapillaris images are exported to Image J software for image processing and calculation of the various parameters of interest (percentage of flow deficit over the entire slice and over the various subsectors).

ELIGIBILITY:
Inclusion Criteria:

* Participant not afflicted by the disease under investigation and without ophthalmological pathology
* Person matched in age (+/- 5 years) and gender to a case (patient with PXE in pre-atrophic stages included in the PXE cohort)
* Signature of informed consent for participation in the protocol
* Adult at time of inclusion Criteria for non-inclusion of research subjects
* Known ophthalmological diseases (maculopathy, glaucoma, optic neuropathy, retinopathy whatever the aetiology)
* Known severe myopia, defined by a sphere > - 6 dioptres
* Diabetic subject
* Unable to carry out the ophthalmological examinations of the study
* Pregnant, breast-feeding or parturient woman
* Person undergoing psychiatric care under constraint
* Person subject to a legal protection measure
* Person not affiliated or not benefiting from a social security scheme

Exclusion Criteria:

* Ophthalmic pathology (maculopathy, glaucoma, optic neuropathy, retinopathy, whatever the etiology) discovered during the ophthalmic workup
* AngioOCT examination inexploitable (artifact and/or image quality less than 50/100 even after pupillary dilation)
* Severe myopia (sphere > - 6 dioptres) discovered during the ophthalmic workup.

Case inclusion critera :

* Patient diagnosed with pseudoxanthoma elasticum, defined according to Plomp's criteria: two out of three features related to PXE: (1) two pathogenic mutations in the ABCC6 gene, and/or (2) disease-specific dermatological changes and/or (3) disease-specific ocular changes;
* Included in the PXE cohort ;
* With pre-atrophic damage, i.e. at least one eye without choroidal neovessels on OCT-A, without previous intravitreal injection of anti-VEGF, and without major retinal atrophy (less than 2 papillary diameters);
* who have had an angiographic OCT (performed during follow-up consultations) with usable results (no artifacts and image quality of 50/100 or better) ;
* patient's non-objection to participation in a study

Case criteria for non-inclusion :

* Other known ophthalmological pathology (maculopathy, glaucoma, optic neuropathy, retinopathy of any etiology)
* Severe myopia, defined by a sphere > - 6 dioptres
* Diabetic subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mean percentage of choriocapillary flow deficits by OCT-A on 6x6 mm scans | Inclusion
  Comparison of macular choriocapillaris flow deficits per OCT angiography (OCT-A) between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage

SECONDARY OUTCOMES:
comparison between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage : - Average percentage of choriocapillaris flow deficits per OCT-A per ETDRS grid sub-sector ; | During inclusion visit
comparison between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage : - Average percentage of choriocapillaris flow deficits per OCT-A per age, over 6x6mm ; | during inclusion visit
comparison between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage : - Average percentage of choriocapillaris flow deficits per OCT-A according to the presence of inflammatory skin lesion in PXE patients ; | During inclusion visit
Average percentage of choriocapillaris flow deficits per OCT-A according to the presence of arterial stenosis of the lower limbs | During inclusion visit
  comparison between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage :
  - Average percentage of choriocapillaris flow deficits per OCT-A according to the presence of arterial stenosis of the lower limbs on Doppler ultrasound in PXE patients ;
Average percentage of choriocapillaris flow deficits per OCT-A according to the presence of carotid artery dysplasia | During inclusion visit
  comparison between healthy controls and patients with pseudoxanthoma elasticum in pre-atrophic stage :
  - Average percentage of choriocapillaris flow deficits per OCT-A according to the presence of carotid artery dysplasia on Doppler ultrasound in PXE patients ;

CONTACTS AND LOCATIONS:
Overall Officials: Laurie MOUROZEAU, Doctor, Principal Investigator — University Hospital, Angers
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Contact investigator principal study and ask sponsor authorization